CLINICAL TRIAL: NCT00871767
Title: An Open-Label, Randomized, 4 Period Crossover, Replicate Study to Assess the Relative Bioavailability of the Phase III and Phase IIb Formulations of AZD5672 in Healthy Male and Female Subjects
Brief Title: AZD5672 Bioavailability Study in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Layton, MD, PhD, Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D1710C00019; EudraCt No. 2009-009423-10
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Rheumatoid Arthritis
Keywords: AZD5672; relative bioavailability; rheumatoid arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — N-(1-(3-(3,5-difluorophenyl)-3-(4-methanesulfonylphenyl)propyl)piperidin-4-yl)-N-ethyl-2-(4-methanesulfonylphenyl)acetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 40 or 100mg AZD5672, Reference formulation
  Interventions: Drug: AZD5672
- 2 (Experimental): 40 or 100mg AZD5672, Test formulation
  Interventions: Drug: AZD5672

INTERVENTIONS:
Drug: AZD5672 — 40 mg tablet (Test formulation)
  Arms: 2
Drug: AZD5672 — 40 mg tablet (Reference formulation)
  Arms: 1
Drug: AZD5672 — 100 mg tablet (Test formulation)
  Arms: 2
Drug: AZD5672 — 100 mg (2 x 50 mg tablet (Reference Formulation)
  Arms: 1

SUMMARY:
The aim of this study is to compare the blood levels achieved with a new formulation of AZD5672 to an existing formulation of AZD5672 used in previous studies

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures
* BMI between 18 and 30 kg/m2
* Medical and surgical history and physical examination without any clinically significant findings
* Non smokers or past smokers who have stopped smoking within the last 6 months.

Exclusion Criteria:

* History of clinically significant cardio- or cerebrovascular, pulmonary, renal, hepatic, neurological, mental or gastrointestinal disorder or any other major disorder that may interfere with the objectives of the study, as judged by the Investigator
* Clinically significant illness as judged by the Investigator, within two weeks before the first administration of investigational product.
* Female subjects who have a positive pregnancy test or who are pregnant or breast-feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-03; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of AZD5672 using PK variables AUC ss and C max ss | Frequent sampling occasions during study periods, with intensive sampling occurring on days 7,14,21 and 28

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | AE assessed throughout whole the study, twice weekly assessment of BP, pulse and safety labs throughout study period

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, Study Chair — AstraZeneca R&D, Alderley Park, UK; Simon Constable, Principal Investigator — ICON Development Solutions, Manchester, UK
Locations (1):
- Research Site, Manchester, United Kingdom